CLINICAL TRIAL: NCT00301067
Title: A Phase I/II Study of High-Dose Calcitriol in Combination With Temozolomide for Patients With Metastatic Melanoma
Brief Title: Phase I/II Study of High-Dose Calcitriol Plus Temodar for Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 05M1; P30CA060553 (NIH); NU-05M1; NU-0310-093; SPRI-NU-05M1
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Melanoma
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Calcitriol; Temozolomide

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design study. (3) patients per dose stratum will be entered in the following cohorts:
  Cohort 1 - Temozolomide and Calcitriol 0.2mcg/kg days 1 + 15
  Cohort 2 - Temozolomide and Calcitriol 0.3 mcg/kg days 1 + 15
  Cohort 3 - Temozolomide and Calcitriol 0.5 mcg/kg days 1 + 15
  Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every 28 day cycle in each cohort.
  If 1 patient experiences dose limiting toxicity (DLT) at any dose, that cohort will be expanded to 6 patients. If 2 patients experience DLT in that cohort, further dose escalation will cease and the cohort immediately preceding that cohort will be considered the maximum tolerated dose (MTD). Alternatively, if no more patients experience DLT, then dose will be escalated to the next cohort.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 - Temozolomide and Calcitriol (Experimental): Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.2 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Interventions: Dietary Supplement: Calcitriol; Drug: Temozolomide
- Cohort 2 - Temozolomide and Calcitriol (Experimental): Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.3 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Interventions: Dietary Supplement: Calcitriol; Drug: Temozolomide
- Cohort 3 - Temozolomide and Calcitriol (Experimental): Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.5 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Interventions: Dietary Supplement: Calcitriol; Drug: Temozolomide
- Expansion - Temozolomide and Calcitriol (Experimental): Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.5 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Interventions: Dietary Supplement: Calcitriol; Drug: Temozolomide

INTERVENTIONS:
Dietary Supplement: Calcitriol — The patient will receive calcitriol in capsule form by mouth on Days 1 and 15 of every cycle
Drug: Temozolomide — The patient will receive temozolomide in capsule form by mouth on Days 2-8 and 16-22 of each 28 study treatment cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Calcitriol may help temozolomide kill more tumor cells by making them more sensitive to the drug. Calcitriol may also stop the growth of melanoma by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the best dose of calcitriol, the side effects of calcitriol when given together with temozolomide, and to see how well they work in treating patients with metastatic stage IV melanoma.

DETAILED DESCRIPTION:
* Phase I: Patients receive oral calcitriol on days 1 and 15 and oral temozolomide on days 2-8 and 16-22. Treatment repeats every 28 days for 2 courses in the absence of unacceptable toxicity. Responding patients continue therapy for up to 6 courses in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of calcitriol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

* Phase II: Patients receive temozolomide and calcitriol at the MTD as in phase I.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant melanoma

  * Any primary tumor site
* Stage IV disease

  * CNS metastases allowed
* Measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension as ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Must have had at least 1 prior systemic therapy
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Patients with no prior systemic therapy are eligible provided they are not candidates for high-dose interleukin-2
* Recovered from all toxic effects of prior therapy
* More than 4 weeks since prior and no concurrent radiotherapy, chemotherapy, or immunotherapy
* More than 4 weeks since prior and no concurrent radiotherapy, chemotherapy, or immunotherapy
* Fertile patients must use effective contraception

Exclusion Criteria:

* Life expectancy less than 4 months
* known HIV positivity
* evidence of active infection requiring antibiotic therapy
* other malignancy within the past 5 years except surgically resected basal cell or squamous cell skin cancer
* significant medical disease which, in the opinion of the investigator, may interfere with study completion
* pregnant or nursing
* Negative pregnancy test
* prior temozolomide or dacarbazine
* investigational agent within 4 weeks prior to study entry
* concurrent magnesium-containing antacids, digitalis, bile-resin binding drugs, or calcium supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01-30 (Actual); Primary Completion 2012-04-05 (Actual); Study Completion 2012-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on January 13, 2005 with an accrual goal of between 19-28 patients. Accrual was suspended on March 22 2007, reopening May 7 2007, suspended again January 4, 2008, reopening February 14 2008 both times for toxicity evaluations. The study closed permanently on October 28, 2011 with 20 patients enrolled on the study.
Groups:
- Cohort 1 - Temozolomide and Calcitriol: Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.2 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Calcitriol: The patient will receive calcitriol in capsule form by mouth on Days 1 and 15 of every cycle
  Temozolomide: The patient will receive temozolomide in capsule form by mouth on Days 2-8 and 16-22 of each 28 study treatment cycle
- Cohort 2 - Temozolomide and Calcitriol: Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.3 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Calcitriol: The patient will receive calcitriol in capsule form by mouth on Days 1 and 15 of every cycle
  Temozolomide: The patient will receive temozolomide in capsule form by mouth on Days 2-8 and 16-22 of each 28 study treatment cycle
- Cohort 3 - Temozolomide and Calcitriol; Expansion - Temozolomide and Calcitriol: Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.5 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Calcitriol: The patient will receive calcitriol in capsule form by mouth on Days 1 and 15 of every cycle
  Temozolomide: The patient will receive temozolomide in capsule form by mouth on Days 2-8 and 16-22 of each 28 study treatment cycle
Period: Completed DLT Period/1st Cycle
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Started | 4 | 3 | 3 | 10 (Patients did not participate in the DLT portion of the trial, they completed 1st cycle of treatment.)
Completed | 3 | 3 | 3 | 9
Not Completed | 1 | 0 | 0 | 1
Not completed — Progressive Disease | 1 | 0 | 0 | 1
Period: Reached 1st Response/2 Cycles
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Started | 3 | 3 | 3 | 9
Completed | 1 | 2 | 2 | 7
Not Completed | 2 | 1 | 1 | 2
Not completed — Progressive Disease | 2 | 1 | 1 | 2
Period: Completed 4 Cycles of Treatment
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Started | 1 | 2 | 2 | 7
Completed | 0 | 1 | 0 | 2
Not Completed | 1 | 1 | 2 | 5
Not completed — Progressive disease | 1 | 1 | 2 | 5
Period: Completed 12 Cycles of Treatment
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Started | 0 | 1 | 0 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 2
Not completed — Progressive Disease | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Follow up Until Death
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Started (All patients that receive treatment on study go into the follow up period for study.) | 4 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2
Not Completed | 1 | 0 | 0 | 1
Not completed — Alive at last data cut point | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Temozolomide and Calcitriol (Cohort 1-3+Expansion): Temozolomide dose of 150 mg/m2 will be administered orally on days 2-8 and 16-22 every cycle where 1 cycle equals 28 days.
  Calcitriol dose of 0.2, 0.3, or 0.5 mcg/kg will be administered orally on days 1 and 15 every cycle where 1 cycle equals 28 days.
  Calcitriol: The patient will receive calcitriol in capsule form by mouth on Days 1 and 15 of every cycle
  Temozolomide: The patient will receive temozolomide in capsule form by mouth on Days 2-8 and 16-22 of each 28 study treatment cycle
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number and Frequency of Dose Limiting Toxicities (DLTs) With High-dose Calcitriol in Combination With Temozolomide
Description: Determine number and frequency of dose limiting toxicities (DLT) of high-dose calcitriol when administered with temozolomide in patients with metastatic melanoma for up to 12 cycles of therapy, where 1 cycle equals 28 days.
  3 patients per dose cohort will be entered into the trial at doses of 0.2, 0.3, and 0.5 mcg/kg of calcitriol administered orally. If 1 patient experiences dose limiting toxicity (DLT) at any dose, that dose cohort will be expanded to a maximum of 6 patients. If 1 additional patient experiences DLT at that dose stratum, further dose escalation will cease and the dose cohort immediately preceding the dose cohort where the 2 experiences of DLT occurred will be considered the MTD. If no additional patients experience DLT, dose escalation to the next higher dose stratum will take place.
  DLT is defined as National Cancer Institute Common Toxicity Criteria, version 3.0 grade 3 toxicity determined to be related to calcitriol.
Time Frame: From start of treatment, up to 12 cycles where 1 cycle equals 28 days
Population: 1 patient enrolled in cohort 1 was not evaluable for this outcome measure as the patient only received 8 days of treatment. Patients enrolled in the expansion cohort were not evaluable for this outcome measure.
Measure: Number; unit: DLT
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol
Number analyzed (Participants) | 3 | 3 | 3
DLT | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Toxicity
Description: Toxicity will be assessed for each patient on a seven-day on/seven-day off temozolomide in combination with high-dose calcitriol for every 2 weeks for up to 12 cycles where 1 cycle equals 28 days. Toxicity will be assessed during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0) and defined by any toxicity determined to be at least possibly related to either study drug (temozolomide or calcitriol).
  In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
  Grade 3 and grade 4 toxicities where relatedness to either study drug could not be ruled out were collected and recorded only.
Time Frame: From the start of treatment and every 2 weeks for a maximum of 12 cycles, and 30 days post last treatment, where 1 cycle equals 28 days
Population: All patients that receive one dose of study drug were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
Number analyzed (Participants) | 4 | 3 | 3 | 9
participants
  Thrombocytopenia | 1 | 0 | 0 | 1
  Vascular | 1 | 0 | 0 | 1
  Nausea | 0 | 0 | 1 | 0
  Vomiting | 0 | 0 | 1 | 0
  Leukopenia | 0 | 0 | 1 | 1
  Fatigue | 0 | 0 | 0 | 1
  Anemia | 0 | 0 | 0 | 2
  Lymphopenia | 0 | 0 | 0 | 2
  Hemorrhage | 0 | 0 | 0 | 1
  Rash | 0 | 0 | 0 | 1
  Anorexia | 0 | 0 | 0 | 1

3. Secondary Outcome: Tumor Response
Description: Determine best tumor response during treatment. Response and progression was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST). The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up.
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: At baseline and every 8 weeks during treatment for a maximum of 12 cycles where one cycle equals 28 days.
Population: Cohort results for this outcome measure are combined as the objective was to determine the tumor response of patients with this drug combination (dose was irrelevant)
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 20
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 1
  Progressive Disease | 17

4. Secondary Outcome: The Relationship Between Vitamin D-receptor Gene Polymorphisms and Tumor Response
Description: Investigate the relationship between vitamin D-receptor (VDR) gene polymorphisms in Taq1 and Fok1 (analyzed from baseline blood sample) and tumor response. VDR gene analysis was completed using PCR-RFLP based assays.
Time Frame: Baseline and at disease progression or when patient goes off study up to a maximum of 12 months
Population: Cohort results for this outcome measure are combined as the objective was to investigate relationship of VDR gene polymorphisms present and tumor response of patients with this drug combination (dose was irrelevant) Data was not collected or analyzed for this outcome measure.
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 0

5. Post Hoc Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) is defined as percentage of patients who's best response to treatment is complete response plus those with partial response.
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From the start of treatment, every 2 cycles where 1 cycle equals 28 days, for a maximum of 12 cycles
Population: Cohort results for this outcome measure are combined as the objective was to determine the ORR of patients with this drug combination (dose was irrelevant)
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 20
Participants | 2

6. Post Hoc Outcome: Time to Progression
Description: Time to progression (TTP) is measured from the start of treatment until the time of first documentation of disease progression.
Time Frame: From the start of treatment, until progressive disease, up to 12 months
Population: Cohort results for this outcome measure are combined as the objective was to determine the TTP for patients with this drug combination (dose was irrelevant)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 20
Months | 1.81 [1.15 to 1.99]

7. Post Hoc Outcome: Overall Survival
Description: Overall Survival (OS) will be measured from first day of treatment until death of any cause. Patients still alive at the last data cut off point will be censored.
Time Frame: From the first day of treatment until death from any cause, up to a maximum of 6 and half years
Population: Cohort results for this outcome measure are combined as the objective was to determine the OS of patients with this drug combination (dose was irrelevant)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 20
Months | 5.5 [2.7 to 12.3]

8. Post Hoc Outcome: Overall Survival (OS) Stratified by Vitamin D-Receptor (VDR) Gene Polymorphisms
Description: Investigate the relationship between vitamin D-receptor (VDR) gene polymorphisms in Taq1 and Fok1 (analyzed from baseline blood sample) and Overall Survival (OS). VDR gene analysis was completed using PCR-RFLP based assays.
Time Frame: at baseline and until death from any cause up to 6 and half years
Population: Cohort results for this outcome measure are combined as the objective was to determine the relationship between VDR gene polymorphisms and OS for patients with this drug combination (dose was irrelevant)
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Temozolomide and Calcitriol (Cohort 1-3+Expansion)
Number analyzed (Participants) | 17
Months
  VDR genotype (tt+/-ff): number analyzed (Participants) | 6
  VDR genotype (tt+/-ff) | 3.8 [2.0 to 5.7]
  non tt+/-ff VDR genotype: number analyzed (Participants) | 11
  non tt+/-ff VDR genotype | 7.4 [3.0 to 12.3]

ADVERSE EVENTS:
Time Frame: Adverse events for the study were collected over a 6 year and 3 month period. For each patient adverse events were collected for a maximum of 12 cycles where 1 cycle equals 28 days.
Arm/Group | Cohort 1 - Temozolomide and Calcitriol | Cohort 2 - Temozolomide and Calcitriol | Cohort 3 - Temozolomide and Calcitriol | Expansion - Temozolomide and Calcitriol
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/3 | 3/3 | 9/10
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 2/3 | 4/10
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Temozolomide and Calcitriol (N=4) | Cohort 2 - Temozolomide and Calcitriol (N=3) | Cohort 3 - Temozolomide and Calcitriol (N=3) | Expansion - Temozolomide and Calcitriol (N=10)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rapidly declining performance status (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slurred speech and drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death related to disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Temozolomide and Calcitriol (N=4) | Cohort 2 - Temozolomide and Calcitriol (N=3) | Cohort 3 - Temozolomide and Calcitriol (N=3) | Expansion - Temozolomide and Calcitriol (N=10)
Anemia (Hemoglobin decrease) (Blood and lymphatic system disorders) | 2 | 2 | 2 | 6
Neutrophils decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytes (white blood count) (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Platelets decreased (thrombocytopenia) (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 6
Fever (General disorders) | 0 | 0 | 1 | 1
Sweating (General disorders) | 1 | 0 | 1 | 0
Weight loss (General disorders) | 0 | 0 | 0 | 5
Weight gain (General disorders) | 0 | 0 | 1 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 2 | 2 | 5
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Dehydration (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 2 | 1 | 9
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 9
Blood in stool (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhage CNS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection NOS (Infections and infestations) | 0 | 0 | 1 | 2
Oral infection (Infections and infestations) | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Limb edema (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Edema in head and neck (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Albumin, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Transaminase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Bicarbonate - low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bilirubin, serum high (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Calcium, serum low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Creatinine - high (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Glucose, serum high (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Lactic acid dehydrogenase (LDH) increase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Sodium, serum low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Confusion (Nervous system disorders) | 0 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Mood alteration - Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Mood alteration - Depression (Psychiatric disorders) | 0 | 1 | 0 | 2
Motor Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 2
Motor Neuropathy - Foot drop (Nervous system disorders) | 1 | 0 | 0 | 0
Lightheadedness (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral vascular accident (CVA) (Nervous system disorders) | 0 | 0 | 0 | 1
Vision changes (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain - NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Menstrual cramps (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 1
Pain not otherwise specified (General disorders) | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No